CLINICAL TRIAL: NCT06224920
Title: Aktivität Von Zerebralen Netzwerken, Amyloid Und Mikroglia Bei Alterung Und Alzheimer-Krankheit
Brief Title: Activity of Cerebral Networks, Amyloid and Microglia in Aging and Alzheimer's Disease
Acronym: ActiGliA
Status: Completed | Type: Observational
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Principal Investigator, Robert Perneczky, principle investigator, Ludwig-Maximilians - University of Munich
Other Study IDs: 17-755 and 17-569
Record Dates: First submitted 2024-01-16; First posted 2024-01-25 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Alzheimer Disease; Corticobasal Syndrome
Keywords: Alzheimer´s disease; corticobasal degeneration; microglial activation; neuroinflammation; amyloid; tau protein
MeSH Terms: conditions — Alzheimer Disease; Corticobasal Degeneration; Neuroinflammatory Diseases; Frontotemporal Dementia | interventions — Magnetic Resonance Imaging; Blood Specimen Collection; Positron-Emission Tomography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Biospecimen collection and processing data is captured by CentraXX (Kairos GmbH, Bochum, Germany), a fully integrated laboratory automation infrastructure. Biological specimens (DNA, RNA, serum, plasma, etc.) are processed in the laboratory using automated equipment (ChemagicStar, decapper/barcode reader and a StarPlus unit, Hamilton Robotics GmbH, Martinsried) and stored at -80 °C in an automated specimen storage and management unit (BIOS M unit, Hamilton Storage GmbH, Bonaduz, Switzerland).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Alzheimer´s disease spectrum: MCI-AD patients Evidence of minor cognitive impairment with essentially preserved everyday competence and evidence of reduced Aβ42 concentration in the cerebrospinal fluid. Score in the CERAD word list 1.5 SD below the normal range.
  Patients with AD-dementia Evidence of pronounced cognitive impairment and relevant impairment of everyday life and evidence of reduced Aβ42 concentration in the cerebrospinal fluid (diagnostic criteria (NIA-AA fulfilled)).
  Interventions: Diagnostic Test: magnetic resonance imaging; Other: electroencephalography; Diagnostic Test: blood and CSF biomarker; Diagnostic Test: positron emission tomography; Diagnostic Test: neuropsychological test
- corticobasal syndrome due to probable 4 repeat taupathy: Evidence of the typical clinical picture of an atypical Parkinson's syndrome with onset of symptoms > 1 year. No evidence of reduced Aβ42 concentration in the cerebrospinal fluid. Fulfillment of the revised Armstrong criteria for probable CBS or the Movement Disorder's Society criteria for suggestive/possible PSP-CBS.
  Interventions: Diagnostic Test: magnetic resonance imaging; Other: electroencephalography; Diagnostic Test: blood and CSF biomarker; Diagnostic Test: positron emission tomography; Diagnostic Test: neuropsychological test
- subjective congnitive decline: Subjective memory impairment, with age-appropriate unremarkable neurocognitive test battery (CERAD) and no evidence of reduced Aβ42 concentration or increased total tau or phospho-tau concentration in the cerebrospinal fluid. Subjective cognitive deterioration over a period of 6 months to 5 years.
  Interventions: Diagnostic Test: magnetic resonance imaging; Other: electroencephalography; Diagnostic Test: blood and CSF biomarker; Diagnostic Test: positron emission tomography; Diagnostic Test: neuropsychological test

INTERVENTIONS:
Diagnostic Test: magnetic resonance imaging — MRI data acquisition was performed on a 3 Tesla MRI scanner with parallel transmission and reception technology (Skyra Magnetom, Siemens Healthcare, Erlangen, Germany). Imaging is performed with a maximum gradient strength of 45mT/m and a maximum slew rate of 200 T/m/s and a 64-element head coil.
Other: electroencephalography — A 20-channel resting EEG (Brain Products, Gilching, Germany) is recorded as part of routine clinical diagnostics in the Department of Psychiatry and Psychotherapy at the LMU to rule out focal neurophysiological pathologies. Within the scope of the present study, an extended examination will be carried out, which includes a 64-channel EEG, including a passive visual paradigm. After completion of the clinical evaluation, the neurophysiological changes in resting activity will be scientifically analyzed in comparison to the MRI and PET data.
  Other Names: eeg
Diagnostic Test: blood and CSF biomarker — Aβ1-42 and 1-40, total tau protein and phosphorylated tau protein 181 (p-Tau), apolipoprotein E (APOE), soluble TREM2 protein, neurofilament light chain and glial fibrillary protein (GFAP) will be determined.
Diagnostic Test: positron emission tomography — According to an established and standardized protocol, PET scans are performed with the TSPO receptor ligand [18F]-GE-180, [18F]flutemetamol for assessment of fibrillar Aβ 162 accumulation and the Tau ligand [18F]-PI-2620. In brief, [18F]GE-180 TSPO PET images (mean dose: 177 ± 17 MBq) with an emission window of 60-80 min after injection will be acquired to measure the activation of glial cells. [18F]Flutemetamol Aβ PET images (average dose: 182 ± 11 MBq) are acquired with an emission window of 90-110 min after injection to assess fibrillar Aβ accumulation. Dynamic [18F]PI-2620 tau PET (average dose: 186 ± 14 MBq) with an emission window of 0-60 minutes after injection are performed for quantification of tau aggregation. Static images of the late phase (20-40 min) are reconstructed. These images are used for further processing and analysis.
  Other Names: PET
Diagnostic Test: neuropsychological test — Trained psychologists at the Memory Clinic of the LMU Hospital administered the CDR, CERAD-NB and Mini-Mental State Examination (MMSE). The CERAD-NB battery was used to generate a total score for the six subscales: semantic fluency (animals/60 s), modified Boston naming test, lexical items, construction practice, lexical items retrieval, and lexical items discrimination, with higher scores indicating better performance.

SUMMARY:
The temporal sequence of microglial activation, changes in functional and structural connectivity and the progression of neurocognitive deficits has not been conclusively clarified. To date, there have been no studies of the topographical and pathogenetic relationship between microglial activation and network degeneration. The main aim of the present study is to investigate the relationships between functional, structural MRI connectivity and microglial activation at different stages of AD in a multimodal approach. Genetic predisposition and biomarkers in blood and cerebrospinal fluid will also be taken into account in order to close the explanatory gap in pathogenesis between the known molecular pathological changes and their effects at system level in an integrative approach.

DETAILED DESCRIPTION:
The main aim of the present study is to investigate correlations between functional and structural MRI connectivity and microglial activation in PET at different stages of AD. Some previous studies have described that especially the brain regions affected by AD-related alterations show increased microglial activity. How these relationships known at the anatomical level relate to changes in functional connectivity is still largely unclear. The multimodal analysis of functional connectivity in the resting networks and the investigation of inflammatory effects using microglia PET may be able to reveal previously unknown neuropathological connections between different stages of AD. Since a direct toxicity effect of Aβ on surrounding neurons can also be assumed, the topography of fibrillar Aβ deposits is also recorded using PET. To date, there are no studies investigating changes in functional and structural connectivity with microglia-associated inflammatory changes and Aβ at different disease stages.

1. evaluation of the correlation of microglial activation determined in PET with the degeneration of functional networks depending on the stage of the disease.

   1. Is microglial activation or Aβ deposition the cause of changes in functional networks?
   2. What is the overlap between microglia- and Aβ-induced network degeneration (modulation of synaptic pruning vs. neurotoxic effect of ß-amyloid)
   3. How reliable is functional connectivity as a biomarker for AD stratification at different disease stages?
   4. What is the temporal and topographical spread of AD pathologies along the hub regions of the resting networks and can a pattern of spread indicative of a specific molecular mechanism be identified?
   5. Does the extent (quantitative and regional) of microglial activation correlate with existing amyloid and tau deposits, as well as network changes? How does microglial activation change in relation to the progression of tau deposits?
2. correlation of inflammatory changes in a multimodal comparison with changes in structural connectivity, metabolic alterations, biomarker abnormalities and changes at the neurotransmitter level.

   1. Is there an image morphologic correlate of soluble TREM2 receptor concentration in cerebrospinal fluid at different disease stages?
   2. What role does oxidative stress (glutathione changes) play in the pathogenesis of AD and is there a connection to other disease-related changes at the multimodal level?
3. are there certain correlations between genetic factors (especially carriers vs. non-carriers of apolipoprotein E, APOE, risk allele ε4 as the strongest genetic risk factor of sporadic AD) and structural or functional connectivity changes depending on the disease stage that can be derived from the multimodal data analysis? a. What is the temporal relationship between microglial activation and Aβ deposits or functional and structural network alterations?

ELIGIBILITY:
Inclusion Criteria:

* Informed consent for the additional examinations, written declaration of consent
* Constant pharmacotherapy in a period of one week before the MRI/EEG/PET examination

Exclusion Criteria:

* Existence of legal guardianship/restricted capacity to consent
* Other severe concomitant psychiatric illnesses, e.g. schizophrenia, bipolar affective disorder
* Clinically relevant depressive symptoms (Beck Depression Inventory, BDI, score > 17/GDS > 5)
* Acute suicidal tendencies
* Drug, medication or alcohol abuse at the time of the study
* Severe traumatic brain injury (> 2nd degree TBI) in the medical history or 1st degree within the last 3 months.
* Evidence of structural damage to the basal ganglia or brainstem
* Severe neurological diseases (such as disc prolapse in the last 6 months, sensory, motor or autonomic polyneuropathies)
* Severe internal diseases (such as manifest arterial hypertension, severe heart disease, pacemaker, respiratory insufficiency)
* Any electronic implants (e.g. pacemakers) or other MRI and/or PET contraindications
* Malignant diseases of any kind in the last 5 years, severe active infectious diseases, chronic and systemic skin diseases
* Bone diseases (such as Paget's disease, osteoporosis with spontaneous fractures, recent fractures)
* Other circumstances which, in the opinion of the investigator, speak against the patient's participation in this study
* Occupational or other radiation exposure >15 mSv/a

Ages: 55 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: recruitment of participants via the outpatient clinics of Department of Psychiatry and Psychotherapy, Department of Neurology and Institute of Stroke and Dementia Research (LMU hospital)
Sampling Method: Non-Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
association of cerebral connectivity with microglia activation patterns | until 06/2024
  association between functional/structural connectivity and TSPO SUVR
Individual regional associations between Aβ-, tau- and neurodegeneration with microglial activation | until 06/2024
  association of regional amyloid and tau with microglial activation (measured by TSPO-PET)
validation of blood-based biomarkers in the differentiation of AD, SCI and CBS cases | until 06/2024
  comparison of AD-related biomarkers (pTau181, Abeta1-42/1-40), plasma apolipoprotein E and inflammatory biomarkers (GFAP, NfL)

IPD SHARING:
Plan to Share IPD: Undecided